CLINICAL TRIAL: NCT03416413
Title: Randomised Controlled Trial of Foam Sclerotherapy Versus Ambulatory Phlebectomy for the Treatment of Varicose Vein Tributaries
Brief Title: Study of Foam Sclerotherapy Versus Ambulatory Phlebectomy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17/WS/0192
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Varicose Veins
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambulatory Phlebectomy (Active Comparator): Ambulatory phlebectomy of varicose vein tributaries
  Interventions: Procedure: Ambulatory phlebectomy
- Foam Sclerotherapy (Active Comparator): Injection of foam sclerosant into varicose vein tributaries
  Interventions: Drug: Foam sclerotherapy

INTERVENTIONS:
Procedure: Ambulatory phlebectomy — Minor surgery to remove varicose vein tributaries
  Arms: Ambulatory Phlebectomy
Drug: Foam sclerotherapy — Injection of foam sclerosant into varicose vein tributaries
  Arms: Foam Sclerotherapy

SUMMARY:
This study will be comparing the treatment of varicose vein tributaries using either foam sclerotherapy or ambulatory phlebectomies. Patients will be randomised to having either ambulatory phlebectomy (group A) or foam sclerotherapy (group B) following treatment of their saphenous vein.

The re-intervention rates, safety, patient experience as well as the cost effectiveness of each intervention will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age
* Symptomatic GSV or SSV vein reflux > 0.5 seconds on colour Duplex
* Varicose vein tributary requiring treatment

Exclusion Criteria:

* Current DVT
* Recurrent varicose veins
* Arterial disease (ABPI<0.8)
* Vein diameter < 3mm
* Preference for one of the treatment options
* Patient who are unwilling to participate
* Inability or unwillingness to complete questionnaires
* Inability to attend follow-up appointments
* Patient currently included in a study of varicose vein treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Re-intervention rate | 12 months
  Re-intervention on varicose vein tributaries during study period

SECONDARY OUTCOMES:
Generic quality of life score | 12 months
  Quality of life score using the EuroQol's EQ-5D [0=worse quality of life; 1=best quality of life]
Disease-specific quality of life score | 12 months
  Quality of life score using the Aberdeen Varicose Vein Questionnaire (AVVQ) [0=worse quality of life; 100= best quality of life]
Disease specific quality of life score | 12 months
  Quality of life score using the ChronIc Venous Insufficiency Quality of Life Questionnaire (CIVIQ) [0=worse quality of life; 100=best quality of life]
Clinical score | 12 months
  Clinical change using the Venous Clinical Severity Score (VCSS) [0=least severe disease; 30=most severe disease]
Clinical score | 12 months
  Using the Clinical-Etiological-Anatomical-Pathophysiological (CEAP) classification [0=no varicose veins; 1=telangiectasia; 2= varicose veins; 3=oedema; 4=skin changes; 5=healed ulcer; 6=ulcer]
Pain score over the first 10 days | 2 weeks
  Pain score over the first 10 days using a 0-100mm visual analogue scale (0=no pain; 100=worst pain)
Degree of bruising at 2 weeks | 2 weeks
  Degree of bruising at 2 weeks using a categorical 0-5 bruising scale (0=no bruising; 5=bruising extending beyond treated segment)
Time to return to normal activities | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Charing Cross Hospital, Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Belramman A, Bootun R, Lane TRA, Davies AH. Foam sclerotherapy versus ambulatory phlebectomy for the treatment of varicose vein tributaries: study protocol for a randomised controlled trial. Trials. 2019 Jul 3;20(1):392. doi: 10.1186/s13063-019-3398-0. PMID 31269978